CLINICAL TRIAL: NCT02788526
Title: The Clinical Randomized Trial of Adjuvant Transarterial Chemo Embolization (TACE) to Reduce the Recurrence in Hepatocellular Carcinoma (HCC) Patients at High Risk After Resection
Brief Title: Adjuvant TACE to Reduce the HCC Recurrence After Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rong-ping Guo, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-HCC-ADTACE
Record Dates: First submitted 2016-03-23; First posted 2016-06-02 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma,Hepatocellular; Chemoembolization; Adjuvant therapy; Hepatocellular; Microvessels invasion
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjuvant TACE (Experimental): Adjuvant TACE were performed 4-6 weeks after surgery
  Interventions: Procedure: Adjuvant TACE
- Follow-up (Other): Routine follow-up were performed instead of adjuvant TACE
  Interventions: Procedure: Follow-up

INTERVENTIONS:
Procedure: Adjuvant TACE — 1~2 cycles TACE were performed as adjuvant therapy after radical hepatectomy
  Arms: Adjuvant TACE
Procedure: Follow-up — Patients received just follow-up to monitor the recurrence of HCC
  Arms: Follow-up

SUMMARY:
Hepatocellular carcinoma (HCC) is the sixth most common malignancies worldwide and the second leading cause of cancer-related death. Surgical resection is still the main radical approach for HCC, but the recurrence rate after hepatectomy is very high, which hampers the further improvement of prognosis of HCC patients. The conventional risk factors of recurrence including: huge tumor, multiple lesions, vessels invasion and tumor rupture. Recently, the microvessels invasion (MVI) has been recognized a novel risk factor of recurrence after hepatectomy. The investigators' previous study showed that the recurrence rate is more than 50% for the patients with >5cm solitary tumor and MVI. The MVI was confirmed as the only independent risk factor for the overall and disease-free survival of HCC patients in multiple variables analysis. It is important to reduce the recurrence and prolong the survival of patients after hepatectomy with effective adjuvant therapy. TACE has been utilized as an adjuvant therapy after hepatectomy, but its significance is still unknown. Then, the investigators design the current prospective randomized clinical trial to evaluate the effect of adjuvant TACE to reduce the recurrence in HCC patients at high risk (>5cm solitary tumor and MVI) after resection, compared to vigilant follow-up.

DETAILED DESCRIPTION:
The patients with solitary tumor more than 5cm and microvessels invasion after radical hepatectomy were randomized to receive adjuvant TACE（1~2 cycles, 4~6 weeks) or follow-up. The main endpoint: overall survival (OS), disease-free survival(DFS), and safety were compared between this two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~75 years;
2. Eastern Cooperative Oncology Group performance status (ECOG PS) score <=2;
3. Histologically confirmed hepatocellular carcinoma with microvessels invasion;
4. No previous treatment for HCC;
5. More than 5 cm solitary tumor before surgery confirmed by more than 2 radiological examinations;
6. R0 resection achieved;
7. No recurrence evidence in radiological follow-up 3~7 weeks after surgery;
8. Adequate hematologic parameters and liver and kidney functions: (1) Neutrophils Absolute >=1.5*10^9/L; (2) Hemoglobin >=90g/L; (3) Platelet count >=75*10^9/L; (4) Serum albumin >=35g/L; (5) Serum total bilirubin <=1.5* upper limit of normal (ULN); (6) Serum Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) <2.5*ULN; (7) Serum creatinine <=1.5*ULN; (8) International normalized ratio (INR) <=1.5;
9. Give signed informed consent before enrollment.

Exclusion Criteria:

1. Function impairment of vital organs (heart, lung, kidney, etc), serious infection or >grade 2 adverse events (Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0);
2. Histologically confirmed of positive resection margin (R1 resection);
3. Previous or current malignant tumor beyond HCC;
4. Allergy to any agent of the TACE regimen;
5. History of organ transplantation;
6. Previously receiving other treatments for HCC;
7. Pregnant or breastfeeding women, and women of childbearing potential without adequate contraception;
8. Neurological or mental abnormalities that may affect cognitive assessment and inform consent;
9. Concomitant anti-tumor therapy or participating in other interventional clinical trials;
10. Other psychological, family or social reason, which would affect compliance with the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years
  The overall survival is defined as the percentage of patients who are alive at 5 years after their enrollments of this study.

SECONDARY OUTCOMES:
Disease-free survival | 5 years
  The disease-free survival is defined as the percentage of patients who are alive at 5 years without any signs or symptoms of HCC after their enrollments of this study.
Safety: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 5 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Rong-ping GUO, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- SUN YAT-SEN University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhong C, Guo RP, Li JQ, Shi M, Wei W, Chen MS, Zhang YQ. A randomized controlled trial of hepatectomy with adjuvant transcatheter arterial chemoembolization versus hepatectomy alone for Stage III A hepatocellular carcinoma. J Cancer Res Clin Oncol. 2009 Oct;135(10):1437-45. doi: 10.1007/s00432-009-0588-2. Epub 2009 May 1. PMID 19408012
- [Background] Li JQ, Zhang YQ, Zhang WZ. [Evaluation of chemoembolization as an adjuvant therapy for primary liver carcinoma after surgical resection]. Zhonghua Zhong Liu Za Zhi. 1994 Sep;16(5):387-9. Chinese. PMID 7895595
- [Background] Li JQ, Zhang YQ, Zhang WZ, Yuan YF, Li GH. Randomized study of chemoembolization as an adjuvant therapy for primary liver carcinoma after hepatectomy. J Cancer Res Clin Oncol. 1995;121(6):364-6. doi: 10.1007/BF01225689. PMID 7541051
- [Background] Peng B, Liang L, He Q, Zhou F, Luo S. Surgical treatment for hepatocellular carcinoma with portal vein tumor thrombus. Hepatogastroenterology. 2006 May-Jun;53(69):415-9. PMID 16795984